CLINICAL TRIAL: NCT03343353
Title: Therapy by Led (Light Emission Diode) in Cutaneous Lesion: in Vivo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor Doctoral, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Therapy led in lesion
Record Dates: First submitted 2017-10-27; First posted 2017-11-17 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Burn Injury
Keywords: burn injury, phototherapy, wound healing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Volunteers will be randomized into groups:
  Group Sham= 35 Group red LED= 35 Group infrared LED = 35
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LED red group (630nm) (Experimental): The leds will initially be measured in the photobiophysics laboratory of the University of São Paulo - Ribeirão Preto, regarding wavelength parameters, beam divergence, nominal power and fluency. The application will be in the graft donor area (scalp) of burn patients. The applied fluence will be 4J / cm2.
  Interventions: Other: LED (Light Emission Diode)
- LED infrared group (940nm) (Experimental): The leds will initially be measured in the photobiophysics laboratory of the University of São Paulo - Ribeirão Preto, regarding wavelength parameters, beam divergence, nominal power and fluency. The application will be in the graft donor area (scalp) of burn patients. The applied fluence will be 4J / cm2.
  Interventions: Other: LED (Light Emission Diode)
- Group Sham (Sham Comparator): This group will not receive irradiation by led light. You will only receive the routine care of the hospital unit to which you are hospitalized. These patients will be evaluated in the same way as the other two intervention groups, and also by a blind evaluator.
  Interventions: Other: LED (Light Emission Diode)

INTERVENTIONS:
Other: LED (Light Emission Diode) — LED light application in cutaneous lesions from the graft donor area (scalp) in patients who are victims of burns

SUMMARY:
Light Emitting Diode (LED) therapy has been investigated in burns and skin ulcers, as it has a bactericidal effect and promotes tissue repair. This study aims to evaluate LED therapy at different wavelengths in the healing process of graft donor area in adult burn victims.

DETAILED DESCRIPTION:
It is a blinded and controlled clinical trial in which burned adult patients will be selected, who will be irradiated with red (630 nm) and infrared (940 nm) LEDs at 4J / cm2 fluency, in the donor area of until complete reepithelialization. Patients included will be the donor scalp area, with withdrawal of 0.2 mm. For application of the LEDs, the device will be calibrated for wavelength parameters, beam divergence, nominal power and fluency in the photobiophysical laboratory of the University of Ribeirão Preto - SP. Three groups will be divided: GS = Sham group (will not receive LED irradiation), will only receive routine hospital care, GT-V = treatment group with red led, and GT-IV = treatment group with infrared led. Patients will be randomized for group distribution. The donor areas will be evaluated by infrared thermography, computerized bioimpedance, infrared plethysmography, and Vancouver healing scale at two times, the first within a period of up to 24 hours after graft surgery, and the second after release of the primary dressing. The evaluations will be carried out by an expert evaluator, blind to the groups. For the analysis of the results will be applied statistical tests intra and intergroup (p <0.05). This research aims to contribute with a new therapeutic method in the control of infections commonly found in cutaneous lesions, as well as in the healing process of the skin.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the Burn Unit of the HCFMRP-USP - Emergency Unit, who agree to participate in the study and are over 18 years of age, guided and without diagnosis of psychiatric diseases, who have undergone graft surgery for a maximum of 24 hours, with a body mass index greater than 16 kg / m² and without infection (sepsis), and that do not present any factor that could interfere in healing such as diabetes or the use of corticosteroids.

Exclusion Criteria: patients who develop infection, are not adherent to treatment or are willing to not continue to participate in the research are excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-02-19 (Estimated); Primary Completion 2020-02-19 (Estimated); Study Completion 2020-02-19 (Estimated)

PRIMARY OUTCOMES:
Detachment of the primary dressing | 2 weeks
  Skin re-epithelialization

SECONDARY OUTCOMES:
The Vancouver Scar Scale (VSS) | 2 weeks
  This scale evaluates the skin in four questions: pigmentation (3 items), vascularization (4 items), malleability (6 items) and scar height (4 itns). It is in the public domain and will be applied by the researcher to evaluate the donor area. Originally developed in the English language by Sullivan et al. (1990), adapted and validated for Portuguese by Santos, Tibola and Marques (2014). The final score varies from 0 to 13, being the lowest score corresponding to the best result (better quality of the scar). The scores are added to each item, and the lower the score, the better the quality of the scar.
Digital Photography | 2 weeks
  Analysis of the size and characteristics of the skin donor area by Image J software
Infrared Thermography | 2 weeks
  Quantitative analysis of skin temperature difference. Skin temperature (Celsius Degree). This evaluation seeks to find possible temperature differences between samples. With precision of up to 0.05 ° C, emissivity of 0.98 will be established, with three infrared images in sequence, and the distance between the thermograph and the donor area will be determined after a pilot test for the scalp regions, thus allowing the best framing and resolution of the area to be evaluated. An infrared thermograph model T400 (FLIR, Wilsonville, United States) will be used.
  The analysis of the images will be by the software QuickReport, version 1.2.
Bioimpedance | 2 weeks
  Analysis of the electrical resistance of the skin donor area. The electrical impedance of the tissue in the healthy skin donor region will be evaluated by the Biodynamics 450® bioimpedance instrument (mark, city, state, country), in which the phase angle in the 50 KHz frequency will be obtained. To do this, prior to the examination, the volunteer will remain in the supine position for 10 minutes, in a room with controlled temperature (22 ± 2ºC) and humidity of 50%. The measurements will be collected by four electrodes that will be coupled 1 cm from the edge of the lesion, for further processing and analysis, being this a relevant parameter to evaluate the effectiveness of the treatment in the process of wound healing (Moore et al., 2011). The impedance between the electrodes will be expressed in kiloohms (KΩ).
Infrared Plesthysmography | 2 weeks
  Changes in the microvascular blood volume of the tissue around the wound

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Flávia Fernanda de Oliveira Assunção, Ribeirão Preto, São Paulo
  - University of Sao Paulo, Ribeirão Preto, São Paulo